CLINICAL TRIAL: NCT05161858
Title: Longitudinal Characterization of Respiratory Tract Exacerbations and Treatment Responses in Primary Ciliary Dyskinesia
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Washington University School of Medicine (Other); Children's Hospital Colorado (Other); Stanford University (Other); Seattle Children's Hospital (Other); The Hospital for Sick Children (Other); McGill University (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 20-0805
Record Dates: First submitted 2021-11-29; First posted 2021-12-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Primary Ciliary Dyskinesia; Kartagener Syndrome
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sputum for inflammatory markers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Primary Ciliary Dyskinesia (PCD) - Well State: Subjects with confirmed PCD in Well State
- Primary Ciliary Dyskinesia (PCD) - Sick State: Subjects with confirmed PCD in Sick State

SUMMARY:
The overall objective of this longitudinal, observational study is to provide information needed to inform the design of future interventional trials of respiratory exacerbation prevention and treatment in children and adults with primary ciliary dyskinesia (PCD).

DETAILED DESCRIPTION:
This is a longitudinal, prospective multicenter study to characterize acute respiratory illnesses (ARIs) and response to treatment in PCD patients. Participants (N=125) will be children age ≥6 years and adults with definite PCD. Participants will be enrolled for approximately 13 months, during which they will attend at least two study visits and perform home monitoring. Participants will be encouraged to attend study visits in-person but will have the option for virtual telehealth visits to ensure compliance with local guidelines and participant safety. Endpoints will be assessed during both well state (i.e., patients typical state of health) and sick state (i.e., during each self-reported period of acute respiratory illness). Informed consent will be obtained, after which the participant will be receive a home spirometer and instructed in its use This design allows for a training period in order to become proficient with home spirometry, with the first study visit occurring 1 month ± 2 weeks after enrollment and the second 12 (±1) months after visit 1 (coordinated with routine clinic visits as possible). Participants will also participate in a set of two optional ARI visits during one ARI, scheduled between 3-5 business days of study team notification by the participant of the new ARI and 2-4 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCD

  1. Clinical features consistent with PCD PLUS
  2. At least 1 diagnostic test consistent with PCD:

  i) Biallelic pathogenic variants in PCD-associated genes identified by genetic panel testing including deletion/duplication analysis; ii) Ciliary ultrastructural defect by transmission electron microscopy known to be disease-causing, including outer dynein arm defects, outer dynein arm plus inner dynein arm (IDA) defects, IDA defects with microtubular disorganization and absent central pair
* Age ≥ 6 years
* At least one course of antibiotics (oral or IV) in the prior year prescribed to treat new or increased respiratory symptoms
* Smart phone and/or internet access available in home
* Informed consent provided by participant or parent/guardian, with assent provided as applicable

Exclusion Criteria:

* Acute course of antibiotics for respiratory symptoms completed <14 days prior to enrollment or Visit 1 (evaluated at enrollment and Visit 1; visit may be rescheduled >14 days after completion of antibiotics)
* Developmental or cognitive disability that would impair ability to complete PRO instruments or perform spirometry
* Congenital heart disease OTHER THAN repaired or resolved atrial septal defect (ASD) or ventricular septal defect (VSD)
* Asplenia or functional asplenia
* Co-existing non-pulmonary disease that, in the opinion of the investigator, could have significant impact on lung function or health-related quality of life (e.g., severe scoliosis) or overall health status (e.g., cancer, severe renal disease)
* Listed for or post-lung transplantation

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects diagnosed with PCD
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Mean FEV1 Percent Predicted Values in Well State and Sick State | 12 months
  Forced expired volume in 1 second (FEV1) will be assessed by percentage of the predicted value (0-100%).
Mean Primary Ciliary Dyskinesia-Quality of Life Score in Well State and Sick State | 12 months
  Domains (scales) include physical, emotional, social, school and role functioning; treatment burden; ears and hearing; upper and lower respiratory symptoms; and vitality. The recall period is one week and responses are rated on a 4-point Likert scale.
Mean PCD-Respiratory Symptom Diary Score Well State and Sick State | 12 months
  The PCD-RSD contains 17 items, 10 on symptoms and 7 on social/emotional impact. The recall period is 24 hours and 15 questions are rated on a 5-point Likert Scale, while two questions are binary (Range: 0-62, 0 being the best and 62 being the worst).

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Rosenfeld, MD, Principal Investigator — Seattle Children's Hospital; Scott Sagel, MD, PhD, Principal Investigator — Children's Hospital Colorado
Locations (7):
- United States (5):
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Washington University in St. Louis, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Seattle Children's Hospital, Seattle, Washington
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
This project is part of the Rare Diseases Clinical Research Network (RDCRN). As such, this project is required to share data with the RDCRN Data Management and Coordinating Center (DMCC) for the purpose of establishing a data repository under National Institutes of Health (NIH) oversight.
Time Frame: The data will become available following the completion of the study and when the DMCC transfers the data to the federal repository.
Access Criteria: • The policies and procedures for requesting and obtaining access to the RDCRN Data Repository will be determined by the NIH program officials responsible for the Data Repository, in consultation with the RDCRN Steering Committee, and will be managed by the RDCRN DMCC.